CLINICAL TRIAL: NCT03449433
Title: A Mixed Meal Tolerance Test Study to Evaluate the Pharmacokinetics and Pharmacodynamics of LY900014 Compared to Humalog Following a Single Dose in Adults With Type 1 Diabetes
Brief Title: A Meal Test Study of LY900014 in Participants With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 16911; I8B-MC-ITSL (Other: Eli Lilly and Company); 2017-003459-47 (EudraCT Number)
Record Dates: First submitted 2018-02-23; First posted 2018-02-28 (Actual); Results first posted 2020-04-30 (Actual); Last update posted 2020-04-30 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- LY900014 (Experimental): T1DM participants received a single, individualized, subcutaneous (SC) dose of LY900014.
  Interventions: Drug: LY900014
- Insulin Lispro (Humalog®) (Active Comparator): T1DM participants received a single, individualized, SC dose of insulin lispro.
  Interventions: Drug: Insulin Lispro
- Insulin Aspart (NovoRapid®) (Active Comparator): T1DM participants received a single, individualized, SC dose of insulin aspart.
  Interventions: Drug: Insulin Aspart
- Insulin Aspart (Fiasp®) (Active Comparator): T1DM participants received a single, individualized, SC dose of insulin aspart.
  Interventions: Drug: Insulin Aspart
- Healthy Participants (No Intervention): Healthy participants who received no study drug.

INTERVENTIONS:
Drug: LY900014 — Administered SC
  Other Names: Ultra-Rapid Lispro
  Arms: LY900014
Drug: Insulin Lispro — Administered SC
  Other Names: Humalog®; LY275585
  Arms: Insulin Lispro (Humalog®)
Drug: Insulin Aspart — Administered SC
  Other Names: NovoRapid®
  Arms: Insulin Aspart (NovoRapid®)
Drug: Insulin Aspart — Administered SC
  Other Names: Fiasp®
  Arms: Insulin Aspart (Fiasp®)

SUMMARY:
Two forms of insulin lispro (LY900014 and Humalog®) and two forms of insulin aspart (NovoRapid® and Fiasp®) will be given to trial participants with diabetes mellitus type 1 by injection under the skin. The study will assess how fast the active ingredient (insulin lispro or insulin aspart) gets into the blood stream and how long it takes the body to remove it. A test meal will be given to trial participants to assess the course of the blood sugar lowering effect of the investigational products. The safety and tolerability of LY900014 will also be assessed. Screening is required within 14 days prior to the lead in. For each participant, the study will last up to 91 days.

ELIGIBILITY:
Inclusion Criteria:

* Are male or female participants with Type 1 Diabetes Mellitus (T1DM) for at least 1 year
* Have a body mass index (BMI) of 18.5 to 35.0 kilogram per meter square (kg/m²)
* Have a glycated hemoglobin (HbA1c) less than (<)9.0 percent (%)
* Have had no episodes of severe hypoglycaemia in the last 6 months

Exclusion Criteria:

- Have a history or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine (apart from T1DM), hematological, or neurological disorders capable of significantly altering the absorption, metabolism or elimination of drugs; of constituting a risk when taking the investigational product; or of interfering with the interpretation of data

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Institut für Stoffwechselforschung, Neuss, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Type 1 Diabetes Mellitus (T1DM) Cohort 1: Period 1: LY900014 administered subcutaneously (SC) immediately before meal Period 2: insulin n Aspart (Fiasp®) administered SC Period 3:Insulin Lispro (Humalog®) administered SC Period 4: Insulin Aspart (NovoRapid®) administered SC
  with 21 hours between doses
- T1DM Cohort 2: Period 1: Insulin Aspart (Fiasp®) administered SC Period 2: LY900014 administered subcutaneously (SC) Period 3: Insulin Aspart (NovoRapid®) administered SC Period 4:Insulin Lispro (Humalog®) administered SC
  with 21 hours between doses
- T1DM Cohort 3: Period 1: Insulin Aspart (NovoRapid®) administered SC Period 2:Insulin Lispro (Humalog®) administered SC Period 3: insulin Aspart (Fiasp®) administered SC Period 4: LY900014 administered subcutaneously (SC)
  with 21 hours between doses
- T1DM Cohort 4: Period 1:Insulin Lispro (Humalog®) administered SC Period 2: Insulin Aspart (NovoRapid®) administered SC Period 3: LY900014 administered SC Period 4: insulin Aspart (Fiasp®) administered SC
  with 21 hours between doses
- Healthy Participants: Healthy participant cohort did not receive any dose of study drug.
Period: Period 1
Arm/Group | Type 1 Diabetes Mellitus (T1DM) Cohort 1 | T1DM Cohort 2 | T1DM Cohort 3 | T1DM Cohort 4 | Healthy Participants
Started | 17 | 16 | 18 | 17 | 12
Received at Least 1 Dose of Study Drug | 17 | 16 | 18 | 17 | 0
Completed | 17 | 16 | 18 | 17 | 12
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Type 1 Diabetes Mellitus (T1DM) Cohort 1 | T1DM Cohort 2 | T1DM Cohort 3 | T1DM Cohort 4 | Healthy Participants
Started | 17 | 16 | 18 | 17 | 12
Received at Least 1 Dose of Study Drug | 17 | 16 | 18 | 17 | 0
Completed | 17 | 16 | 18 | 17 | 12
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Type 1 Diabetes Mellitus (T1DM) Cohort 1 | T1DM Cohort 2 | T1DM Cohort 3 | T1DM Cohort 4 | Healthy Participants
Started | 17 | 16 | 18 | 17 | 12
Received at Least 1 Dose of Study Drug | 17 | 15 | 18 | 17 | 0
Completed | 17 | 15 | 18 | 17 | 12
Not Completed | 0 | 1 | 0 | 0 | 0
Period: Period 4
Arm/Group | Type 1 Diabetes Mellitus (T1DM) Cohort 1 | T1DM Cohort 2 | T1DM Cohort 3 | T1DM Cohort 4 | Healthy Participants
Started | 17 | 15 | 18 | 17 | 12
Received at Least 1 Dose of Study Drug | 17 | 15 | 18 | 17 | 0
Completed | 17 | 15 | 18 | 17 | 12
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants that received at least 1 dose of study drug.
Groups:
- T1DM Cohort: All randomized participants with T1DM participants who received at least 1 dose of study drug.
- Healthy Participants: All healthy participants.
- Total: Total of all reporting groups
Arm/Group | T1DM Cohort | Healthy Participants | Total
Number analyzed (Participants) | 68 | 12 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 12 | 73
  >=65 years | 7 | 0 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 0 | 17
  Male | 51 | 12 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 67 | 12 | 79
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 68 | 12 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 68 | 12 | 0
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per meter squared] | 25.82 (2.36) | 25.38 (1.80) | 25.38 (1.80)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Insulin Lispro or Insulin Aspart Area Under the Concentration Curve From Zero to Seven Hours (AUC 0-7h) Following Administration of Each Study Arm
Description: PK: Insulin Lispro or Insulin Aspart AUC(0-7h)
Time Frame: 0 (predose), 1, 2, 3,5,10, 15, 20, 25, 30,35, 40, 45, 50, 55,60, 70, 90, 120, 150,180, 240, 300, 360 and 420 minutes postdose
Population: All randomized, T1DM participants who received at least 1 dose of study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomols times hour per Liter
Groups:
- Insulin Lispro (Humalog®): T1DM participants received a single,individualized, SC dose of insulin lispro (Humalog)
- Insulin Aspart (NovoRapid®): T1DM participants received a single,individualized, SC dose of insulin
- Insulin Aspart (Fiasp®): T1DM participants received a single,individualized, SC dose of insulin aspart
Arm/Group | LY900014 | Insulin Lispro (Humalog®) | Insulin Aspart (NovoRapid®) | Insulin Aspart (Fiasp®)
Number analyzed (Participants) | 62 | 62 | 62 | 62
picomols times hour per Liter | 786 (36) | 756 (37) | 938 (41) | 928 (36)
Statistical Analysis 1: Comparison: LY900014 vs Insulin Lispro (Humalog®); Test type: Superiority; Ratio of LS Means = 1.04, 95% CI 2-sided [0.985 to 1.10]

2. Secondary Outcome: Pharmacodynamics (PD): Change From Baseline Area Under the Concentration Curve of Glucose Relative to a Mixed Meal Tolerance Test (MMTT)
Description: PD: AUC(0-5h) of Glucose Relative to a Mixed Meal Tolerance Test (MMTT)
Time Frame: Time Frame:-30, -15, 0 (predose), 10, 20, 30, 40, 50, 60, 70, 80, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 225, 240, and 300 minutes postdose
Population: All randomized participants who evaluable PD parameters.
Measure: Mean (Standard Deviation); unit: milligrams times hour per deciliter
Groups:
- Insulin Lispro (Humalog®): T1DM participants received a single,individualized, SC dose of insulin lispro (Humalog®) T1DM participants
- Insulin Aspart (NovoRapid®); Insulin Aspart (Fiasp®): T1DM participants received a single,individualized, SC dose of insulin aspart
- Healthy Participants: Healthy participants, cohort did not receive study drug.
Arm/Group | LY900014 | Insulin Lispro (Humalog®) | Insulin Aspart (NovoRapid®) | Insulin Aspart (Fiasp®) | Healthy Participants
Number analyzed (Participants) | 67 | 67 | 67 | 67 | 12
milligrams times hour per deciliter | 81.5 (212) | 141 (224) | 157 (243) | 101 (226) | 44.1 (32.5)

ADVERSE EVENTS:
Time Frame: up to 6 weeks
Groups:
- LY900014: T1DM participants received a single, subcutaneous (SC) dose of LY900014.
- Insulin Lispro (Humalog®): T1DM participants received a single, SC dose of insulin lispro (Humalog®).
- Insulin Aspart (Fiasp®): T1DM participants received a single, SC dose of insulin aspart (Fiasp®).
- Insulin Aspart (NovoRapid®): T1DM participants received a single, SC dose of insulin aspart (NovoRapid®).
- Healthy Participants: Healthy subject cohort, cohort did not receive any dose of study drug.
Arm/Group | LY900014 | Insulin Lispro (Humalog®) | Insulin Aspart (Fiasp®) | Insulin Aspart (NovoRapid®) | Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/67 | 0/68 | 0/67 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 0/68 | 0/67 | 0/12
Other Adverse Events (participants affected / at risk) | 0/68 | 0/67 | 0/68 | 0/67 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-04-10): https://cdn.clinicaltrials.gov/large-docs/33/NCT03449433/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/33/NCT03449433/SAP_001.pdf